CLINICAL TRIAL: NCT06618105
Title: A Prospective, Randomized, Single-dose, Double-blind, Double-dummy, Four-period, Four-treatment Crossover Pivotal Bronchoprovocation Study to Demonstrate the Pharmacodynamic Bioequivalence of Albuterol Sulfate HFA Inhalation Aerosol (E.Q. 90 mcg of Albuterol Base/Inh) (of Macleods Pharmaceuticals Ltd.) to Albuterol Sulfate HFA Inhalation Aerosol (E.Q. 90 mcg of Albuterol Base/Inh) (Distributed by Teva Pharmaceuticals USA, Inc.) in Adult Patients With Stable Mild Asthma
Brief Title: Bronchoprovocation Study to Demonstrate the Pharmacodynamic Bioequivalence of Albuterol Sulfate HFA Inhalation Aerosol (E.Q. 90 mcg of Albuterol Base/Inh) of Macleods Pharmaceuticals Ltd
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Macleods Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-060-ALBU-2024; Bio-IND #172701 (Other: U.S. Food and Drug Administration)
Record Dates: First submitted 2024-09-17; First posted 2024-10-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Mild Asthma
Keywords: Bronchoprovocation Study
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Single-dose, Double-blind, Double-dummy, Four-period, Four-treatment Crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Zero dose (Placebo) (Placebo Comparator): One actuation (oral inhalation) each from two different placebo R inhalation aerosols and one actuation (oral inhalation) each from two different placebo T inhalation aerosols
  Interventions: Drug: Test Placebo; Drug: Reference Placebo
- E.Q. 90 mcg Base dose of R inhalation aerosol (Active Comparator): One actuation (oral inhalation) each from the R inhalation aerosol and the placebo R inhalation aerosol and one actuation (oral inhalation) each from two different placebo T inhalation aerosols
  Interventions: Drug: Test Placebo; Drug: Reference Placebo; Drug: Albuterol Sulfate 90 MCG/INHAL Metered Dose Inhaler, 200 Actuations
- E.Q. 180 mcg Base dose of R inhalation aerosol (Active Comparator): One actuation (oral inhalation) each from two different R inhalation aerosols and one actuation (oral inhalation) each from two different placebo T inhalation aerosols
  Interventions: Drug: Test Placebo; Drug: Albuterol Sulfate 90 MCG/INHAL Metered Dose Inhaler, 200 Actuations
- E.Q. 90 mcg Base dose of T inhalation aerosol (Experimental): One actuation (oral inhalation) each from the T inhalation aerosol and the placebo T inhalation aerosol and One actuation (oral inhalation) each from two different placebo R inhalation aerosols
  Interventions: Drug: Albuterol Sulfate 90 MCG/INHAL Metered Dose Inhaler, 200 Actuations; Drug: Test Placebo; Drug: Reference Placebo

INTERVENTIONS:
Drug: Albuterol Sulfate 90 MCG/INHAL Metered Dose Inhaler, 200 Actuations — Albuterol sulfate HFA Inhalation Aerosol (E.Q. 90 mcg of albuterol Base/Inh) (of Macleods Pharmaceuticals Ltd.)
  Other Names: Albuterol Sulfate
  Arms: E.Q. 90 mcg Base dose of T inhalation aerosol
Drug: Test Placebo — Matching Placebo of T inhalation aerosol
  Other Names: Placebo
Drug: Reference Placebo — Matching Placebo of R inhalation aerosol
  Other Names: Placebo
  Arms: E.Q. 90 mcg Base dose of R inhalation aerosol; E.Q. 90 mcg Base dose of T inhalation aerosol; Zero dose (Placebo)
Drug: Albuterol Sulfate 90 MCG/INHAL Metered Dose Inhaler, 200 Actuations — Albuterol sulfate HFA Inhalation Aerosol (E.Q. 90 mcg of albuterol Base/Inh) (distributed by Teva Pharmaceuticals USA, Inc.)
  Other Names: Albuterol Sulfate
  Arms: E.Q. 180 mcg Base dose of R inhalation aerosol; E.Q. 90 mcg Base dose of R inhalation aerosol

SUMMARY:
This is a pharmacodynamic bioequivalence bronchoprovocation study using single-dose, double-blind, double-dummy, randomized, study consisting of four study treatments (zero dose [Placebo], E.Q. 90 mcg Base dose of R inhalation aerosol, E.Q. 180 mcg Base dose of R inhalation aerosol, E.Q. 90 mcg Base dose of T inhalation aerosol) and four Periods (Period 1 to Period 4). Randomization procedure at Period 1 will assign any one study treatment to be administered in each Period in a cross-over manner. By the end of Period 4, a subject who completes dosing in all four Periods would have administered all four treatments in the study.

The efficacy variable, post-dose PC20 obtained during each Period is the provocative concentration of the methacholine challenge agent required to reduce the FEV1 by 20% following administration of differing doses of albuterol (or placebo) by inhalation. The 20% reduction in FEV1 is determined as compared to post-saline FEV1 measured before the Placebo or Albuterol administration.

The pharmacodynamic equivalence will be based on the dose-scale method of analysis of the post-dose PC20 If the 90% confidence interval for the relative bioavailability (F) falls within 67.00% -150.00% then it will be considered that pharmacodynamic equivalence is established.

DETAILED DESCRIPTION:
The study consists of screening period (up to 10 days) and four study treatments/ study treatment periods (Period 1, Period 2, Period 3, and Period 4) and a telephonic contact on 2nd day (±1 day) after Period 4 dosing day/last dose of study treatment.

To participate in the study, every subject must provide a signed written informed consent. After obtaining consent subject's eligibility to participate in the study will be confirmed during the screening period.

The study involves bronchoprovocation study using methacholine as challenge agent. Therefore a methacholine challenge test (MCT) will be conducted during screening and at each Period. A MCT involves four steps; Step 1 to Step 4.

In Step 1 (Pre-challenge): Pre-saline/Baseline spirometry will be conducted In Step 2 (saline): saline control test and spirometry: Subjects will be nebulized with normal saline for 1 minute by tidal breathing method. FEV1 will be obtained at about 30 seconds and 90 seconds post-nebulization.

In Step 3 (challenge) methacholine administration and spirometry: Subjects will be nebulized with doubling concentrations of methacholine for 1 minute. Nebulization will start from the lowest methacholine concentration followed by higher doubling concentration until FEV1 value reduces more than or equal to 20% relative to post-saline FEV1 or the highest methacholine concentration is administered or subject is clinically unstable (whichever comes first). After each concentration is nebulized, subject's heart rate will be measured using pulse oximeter and well-being will be checked. FEV1 will be obtained at about 30 seconds and 90 seconds post-nebulization of each methacholine concentration. FEV1 maneuver should meet the acceptability criteria. Each FEV1 will be checked for 20% fall relative to FEV1 obtained in Step 2.

In Step 4 (subject recovery and spirometry): Oral inhalations of recovery medication (Albuterol HFA inhalation aerosol [E.Q. 90 mcg albuterol base/inh]) will be administered to expedite the return of the FEV1 within 90% of FEV1 obtained in Step 1.

During the study Screening-MCT A will be conducted to assess airway responsiveness to methacholine demonstrated by pre-albuterol dose (baseline/Scr-MCTA) PC20 ≤1.56 mg/mL.

Screening-MCT B will be conducted to assess airway responsiveness to methacholine demonstrated by post-two-albuterol-doses (Albuterol HFA inhalation aerosol [90 mcg of albuterol base/inh] Period MCT will be conducted to obtain post-dose PC20 for the primary endpoint. Study treatment dosing will be administered after Step 2 is completed and before initiation of Step 3. Subjects will administer one oral inhalation from four different inhalers with one minute interval between each oral inhalation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant, non-lactating female subjects aged between 18 to 65 years (both ages inclusive)
2. Stable mild asthmatics based on National Asthma Education and Prevention Programme (NAEPP) guidelines
3. Subjects who were diagnosed by physician with mild asthma at least 6 months prior to screening visit date
4. Pre-bronchodilator forced expiratory volume in one second (FEV1) ≥ 80% of predicted
5. Airway responsiveness to methacholine demonstrated by pre-albuterol-dose (baseline) PC20 less than or equal to 1.56 mg/mL using AeroEclipse II BAN and 1-minute tidal breathing method at Screening MCT A
6. The ≥20% reduction in FEV1 at Screening MCT A relative to post-saline FEV1 should be obtained above the lowest methacholine concentration
7. At Screening MCT-B, subjects should have at least four-fold increase in PC20 over Screening MCT-A
8. At Screening MCT -B, the ≥ 20% reduction in FEV1 relative to post saline FEV1 must be obtained up to methacholine concentration 24.96 mg/mL
9. Non-smokers for at least six months prior to screening visit and a maximum smoking history of five-pack years (the equivalent of one pack per day for five years)
10. Women of child-bearing potential or women who are less than or equal to 1 year postmenopausal prior to screening visit must have negative result for urine pregnancy test
11. Women of child-bearing potential or women who are less than or equal to 1 year postmenopausal prior to screening visit must agree to the use of a reliable and medically acceptable method of contraception throughout the duration of the study
12. Women of child-bearing potential or women who are less than or equal to 1 year postmenopausal prior to screening visit using hormonal contraception must be on the same hormonal contraceptive for at least thirty days before the screening period and must be continued same throughout the study.
13. Able to provide signed written informed consent and willing to comply with all aspects of the clinical study protocol

Exclusion Criteria:

* 1.Subjects with FEV1 < 1.5L during methacholine challenge test 2.Evidence of upper or lower respiratory tract infection (e.g., pneumonia, bronchitis, sinusitis) within six weeks prior to the study.

  3.History of seasonal asthma exacerbations, in which case the subject should be studied outside of the relevant allergen season 4.History of cystic fibrosis, bronchiectasis or other respiratory diseases other than asthma (e.g., COPD, interstitial lung disease) 5.Treatment in an emergency room or hospitalization for acute asthmatic symptoms within past three months prior to screening visit 6.Need for daily oral corticosteroids within past three months prior to screening visit 7.History of life-threatening asthma leading to hospitalization within the past 1 year prior to screening visit 8.Known intolerance or hypersensitivity to any component of the albuterol metered dose inhaler (MDI) 9.Uncontrolled hypertension (systolic BP >200 mmHg, or diastolic BP >100 mmHg) 10.History or evidence of myocardial infarction or stroke 11.History of known aortic aneurysm 12.Current use of cholinesterase inhibitor medication (for myasthenia gravis) 13.Clinically significant ECG recording at screening such as flattening of T wave, prolongation of QTc interval (>450 milliseconds), and ST segment depression, which in the opinion of the Investigator, would compromise subject's safety or interfere with the study results 14.History of recent eye surgery or intracranial pressure elevation risk 15.Uncontrolled diabetes (HbA1c ≥9%) at screening 16.Evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled artery disease, cardiac dysrhythmia, or ECG with evidence of ischemic heart disease. In addition, historical or current evidence of significant hematologic, hepatic neurologic, psychiatric, renal, or other disease or that, in the opinion of the Investigator, would put the subject at risk through study participation, or would affect the study analyses if the disease exacerbates in the study 17.Presence of any abnormal clinically significant laboratory investigation at screening visit 18.History of paradoxical bronchospasm 19.Has participated in another investigational study or device research study within 30 days before screening visit date 20.Women are pregnant, breast-feeding, or planning pregnancy during study

Period continuation criteria If subject does not meet any one Period continuation criteria at any visit of Period; retest visit will be conducted and study treatment dosing should not be administered. Period continuation criteria will be checked for maximum three visits.

If subject does not meet all Period continuation criteria at any one visit and within three consecutive visits:

At Period 1: subject should not be randomized and will be considered a 'randomization failure' At Period 2 to Period 4: subject should not administer study treatment dosing and must be discontinued from the study

1. Baseline FEV1 should not be less than 70% of predicted normal value and should be within 88 -112% of qualifying day FEV1 value.

   Baseline FEV1: highest pre-saline FEV1 obtained prior to saline control test at Period MCT and which has met the acceptability criteria and have repeatable quality grade A, B, C mentioned in ATS 2019 standards Qualifying day FEV1 value: highest pre-saline FEV1 obtained prior to saline control test on qualifying day and which has met the acceptability criteria and have repeatable quality grade A, B, C mentioned in ATS 2019 standards and which has not met the retest criteria for Scr-MCT A on qualifying day

   -Qualifying day: Scr-MCT A PC20 is obtained and the results of the Scr-MCT A on this day confirms that subject has met inclusion criteria 4, 5, and 6
2. Baseline FEV1 should be ≥ 1.5 L
3. Baseline FEV1 should meet FEV1 acceptability criteria as mentioned in ATS 2019 standards
4. Baseline FEV1 should meet repeatability quality grade A, B, or C as mentioned in ATS 2019 standards
5. Fall in FEV1 due to the saline control (i.e. post-saline FEV1) should not be more than 10% from the baseline FEV1 Post-saline FEV1: is the highest post-saline FEV1 value from at least one acceptable FEV1 maneuver obtained after nebulization with normal saline is completed (i.e. after saline control test is completed)
6. At least one FEV1 obtained after saline control test (post-saline FEV1) should meet acceptability criteria mentioned in ATS 2019 standards

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Post-dose PC20 (MG/ML) | Post-dose following single-dose administration of differing doses of albuterol or placebo by inhalation, a total of approximately 5 weeks.
  * PC20 which is the provocative concentration of the methacholine challenge agent required to reduce the FEV1 by 20% following administration of differing doses of albuterol (or placebo) by inhalation
  * The 20% reduction in FEV1 is determined as compared to post-saline FEV1 measured before the Placebo or Albuterol administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Multiple Locations, India

IPD SHARING:
Plan to Share IPD: No